CLINICAL TRIAL: NCT01184001
Title: A Phase 1, Randomized, 2-Period, 2-Sequence, Open Label, Single Dose, Cross-Over Study To Evaluate The Effect Of Food On Pharmacokinetics Of Tasocitinib (CP-690,550) Tablets In Healthy Subjects
Brief Title: A Study To Evaluate The Effect Of Food On How Tasocitinib (CP-690,550) Is Absorbed And Moves Through The Body Following Oral Administration Of Tasocitinib (CP-690,550) Tablets To Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A3921076
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Healthy subjects; Food Effect Study
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental)
  Interventions: Drug: Treatment A; Drug: Treatment B
- Sequence 2 (Experimental)
  Interventions: Drug: Treatment B; Drug: Treatment A

INTERVENTIONS:
Drug: Treatment A — Single dose of tasocitinib (CP-690,550) 10 mg under fed conditions.
  Arms: Sequence 1
Drug: Treatment B — Single dose of tasocitinib (CP-690,550) 10 mg under fasted conditions.
  Arms: Sequence 1
Drug: Treatment B — Single dose of tasocitinib (CP-690,550) 10 mg under fasted conditions.
  Arms: Sequence 2
Drug: Treatment A — Single dose of tasocitinib (CP-690,550) 10 mg under fed conditions.
  Arms: Sequence 2

SUMMARY:
In this study, a 10 mg tasocitinib (CP-690,550) tablet will be administered to healthy subjects on two separate dosing occasions. On one occasion the tasocitinib (CP-690,550) tablet will be administered in a fasting condition; On the other occasion the tasocitinib (CP-690,550) tablet will be administered in a fed condition following a standard breakfast meal. The amount of tasocitinib (CP-690,550) in the blood will be measured at various times over 24 hours following each dosing occasion and compared to evaluate for any differences.

DETAILED DESCRIPTION:
To evaluate the effect of food on the pharmacokinetics of tasocitinib (CP-690,550).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-childbearing potential) subjects between the ages of 21 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight for males>50 kg (110 lbs). For females, total body weight >45 kg (99 lbs).
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)

Exclusion Criteria:

* Evidence or history of any clinically significant illness, medical condition, or disease.
* Evidence or history of any clinically significant infections within the past 3 months.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
AUCinf and Cmax of tasocitinib (CP-690,550). | PK blood samples out to 24 hours post dose in each of two periods.

SECONDARY OUTCOMES:
AUClast, Tmax, and t1/2 of tasocitinib (CP-690,550). | PK blood samples out to 24 hours post dose in each of two periods.
Safety: Laboratory tests. | Pre-dose on Day O of Period 1 and post-dose on Day 2 of Period 2.
Safety:Vital signs. | Prior to dosing in Period 1 and 2.
Safety: AE reporting. | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921076&StudyName=A%20Study%20To%20Evaluate%20The%20Effect%20Of%20Food%20On%20How%20Tasocitinib%20%28CP-690%2C550%29%20Is%20Absorbed%20And%20Moves%20Through%20The%20Body%20Following%20Oral%20A